CLINICAL TRIAL: NCT04939467
Title: A Phase 1, Open-Label, Non-Randomized, Fixed Sequence Study to Evaluate the Steady-state Pharmacokinetics of BLD-0409, Nintedanib and Pirfenidone When Administered Concurrently in Healthy Volunteers
Brief Title: Dedicated Drug-Drug Interaction (DDI) Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Blade Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: B-0409-104
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Drug Drug Interaction
MeSH Terms: interventions — pirfenidone; Tablets; nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pirfenidone & BLD-0409 (Experimental): Following an overnight fast, subjects will be administered IP in a fixed sequence.
  Interventions: Drug: Pirfenidone 267 mg Oral Tablet; Drug: BLD-0409 750 mg Oral Tablet
- Nintedanib & BLD-0409 (Experimental): Following an overnight fast, subjects will be administered IP in a fixed sequence.
  Interventions: Drug: Nintedanib 150 mg Oral Capsule; Drug: BLD-0409 750 mg Oral Tablet

INTERVENTIONS:
Drug: Pirfenidone 267 mg Oral Tablet — Fixed sequence use of active product, TID
  Arms: Pirfenidone & BLD-0409
Drug: Nintedanib 150 mg Oral Capsule — Fixed sequence use of active product, BID
  Arms: Nintedanib & BLD-0409
Drug: BLD-0409 750 mg Oral Tablet — Fixed sequence use of active product, QD

SUMMARY:
A Phase 1, Open-Label, Non-Randomized, Fixed Sequence Study to Evaluate the Steady-state Pharmacokinetics of BLD-0409, Nintedanib and Pirfenidone when Administered Concurrently in Healthy Volunteers

DETAILED DESCRIPTION:
This is a single-center, open-label study designed to determine the effect of BLD-0409 on the PK of nintedanib and pirfenidone, all at steady state, and to evaluate the safety and tolerability of BLD-0409 administered with either nintedanib or pirfenidone in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants 18-55 years of age (inclusive) at the time of signing the ICF.
2. Participants must be in good general health, in the opinion of the investigator, with no significant medical history, have no clinically significant abnormalities on physical examination at Screening, and/or before administration of the initial dose of IP.
3. Participants must have clinical laboratory values within normal ranges or < 1.2 times upper limit of normal (ULN) as specified by the testing laboratory, unless deemed not clinically significant (NCS) by the investigator.
4. Body mass index (BMI) 18 to ≤ 30 kg/m2.
5. Female participants must use double barrier contraception and refrain from oocyte donation from at least 28 days prior to Screening and for 90 days after last dose of IP.
6. Male participants and female partners of male participants must agree to use highly effective, double barrier contraception and refrain from sperm donation from first dose of IP and for 90 days after last dose of IP.
7. Females of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day -1. Females not of childbearing potential must be surgically infertile or post-menopausal (defined as cessation of regular menstrual periods for at least 12 months), confirmed by follicle-stimulating hormone (FSH) level >40 mIU/mL at Screening.
8. Participants must provide signed informed consent prior to study entry and have the ability and willingness to attend and comply with the necessary visits at the study site.

Exclusion Criteria:

1. Recent (less than 6 weeks) wound, or presence of an ongoing non-healing skin wound.
2. Presence of any underlying physical or psychological medical condition that, in the opinion of the investigator, would make it unlikely that the participant will complete the study per protocol.
3. Known cardiac disease.
4. Active malignancy and/or history of malignancy in the past 5 years, with the exception of completely excised non-melanoma skin cancer or low grade cervical intraepithelial neoplasia.
5. Serious local or systemic infection within 1 month of Screening requiring antibiotic treatment or history of recurrent infections.
6. Any acute illness within 30 days prior to Day 1.
7. Surgery, bone fracture or major musculoskeletal injury within the past 3 months prior to the first IP administration determined by the investigator to be clinically relevant.
8. Positive for human immunodeficiency virus (HIV) antibody or antigen.
9. Positive hepatitis C virus (HCV) antibody or positive hepatitis B surface antigen (HBsAg).
10. Systolic blood pressure (BP) > 150 mmHg or < 90 mmHg or diastolic BP >90 mmHg or <50 mmHg at Screening with one repeat allowed per the investigator's discretion at Screening and Day -1.
11. Heart rate < 40 beats per minute (bpm) or > 100 bpm at Screening.
12. Prolonged QT interval corrected by Fridericia's formula (QTcF) (>450 ms for males and >470 ms for females), cardiac arrhythmia, or any clinically significant abnormality in the resting ECG, as judged by the investigator.
13. All prescription and over-the-counter medications (including herbal medications), except for contraceptives, are prohibited within 7 days prior to the first IP administration and throughout the entire duration of the study.
14. All vaccines within 14 days prior to first IP administration and throughout the entire duration of the study.
15. Administration of investigational product in another study within 30 days prior to the first IP administration (except BLD-0409), or five half-lives, whichever is longer.
16. Significant weight loss or gain between Screening and first IP administration.
17. Blood donation or significant blood loss within 60 days prior to the first IP administration.
18. Plasma donation within 7 days prior to the first IP administration.
19. Females who are pregnant or breastfeeding.
20. Diets that could alter metabolism (i.e., high protein, Slim Fast®, Nutrisystem®, etc.) within 7 days prior first IP administration.
21. History or presence of alcohol or drug abuse within the 1 year prior to the first IP administration, and unwillingness to be totally abstinent during the treatment period.
22. Positive urine drug screen/alcohol breath test at Day -1 (admission). Repeat urine drug screens will be permitted for suspected false positive results.
23. Intake of alcohol or caffeine-containing products from 48 hours before first IP administration through the EOS visit.
24. Active smokers and users of nicotine-containing products. Note, participants must discontinue smoking/use of nicotine-containing products from 48 hours before first IP administration through the EOS visit.
25. Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Maximum observed drug concentration (Cmax) | Up to 18 days
  Estimated from plasma concentration
Time of the maximum drug concentration (Tmax) | Up to 18 days
  Estimated from plasma concentration
Area under the drug concentration-time curve (AUC) as follows: Pirfenidone - AUC0-8 (Arm 1); Nintedanib - AUC0-12 (Arm 2); BLD-0409 - AUC0-24 (both arms). | Up to 18 days
  Estimated from plasma concentration

SECONDARY OUTCOMES:
Incidence, nature and severity of treatment-emergent adverse events (TEAEs) and Serious Adverse Events (SAEs) | Up to 18 days
  Safety and tolerability will be assessed based on the incidence, nature and severity of TEAEs and SAEs, and changes in safety laboratories, vitals and ECGs

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly S Cruz, MD, Principal Investigator — Advanced Pharma CR, LLC
Locations (1):
- Advanced Pharma, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No